CLINICAL TRIAL: NCT03074292
Title: Comparison Between Effect of Conventional, Intensive and Light Emitting Diodes (LED) Phototherapy on Oxidative Stress Among Neonates With Unconjugated Hyperbilirubinemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rania Ali El-Farrash (Other)
Responsible Party: Sponsor-Investigator, Rania Ali El-Farrash, Assistant professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 00006444
Record Dates: First submitted 2017-02-16; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Oxidative Stress; Neonatal Hyperbilirubinemia; Phototherapy Complication
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- conventional phototherapy (Active Comparator): neonates with unconjugated hyperbilirubinemia exposed to conventional phototherapy
  Interventions: Procedure: phototherapy
- extensive phototherapy (Active Comparator): neonates with unconjugated hyperbilirubinemia exposed to extensive phototherapy
  Interventions: Procedure: phototherapy
- LED phototherapy (Active Comparator): neonates with unconjugated hyperbilirubinemia exposed to LED phototherapy
  Interventions: Procedure: phototherapy

INTERVENTIONS:
Procedure: phototherapy — estimate oxidative stress and trace elements in neonates with unconjugated hyperbilirubinemia after exposure to phototherapy

SUMMARY:
The aim of the present study is to test a hypothesis assuming that phototherapy might have an effect on oxidant/antioxidant status in term and late-preterm neonates with unconjugated hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

* Term and late-preterm neonates (≥35weeks) according to the guidelines of the American Academy of Pediatrics (2004) which stated that gestational ages of newborns were determined according to the first day of the mother's last menstrual period (by the mother's statement) and were additionally confirmed by the Ballard scoring system (Ballard et al., 1991) and antenatal ultrasonographic estimation or obstetric records if present.
* Clinical significant indirect hyperbilirubinemia requiring phototherapy in the first week of life.
* Normal blood counts and peripheral blood smears
* Normal reticulocytic count.
* Breast fed newborn.

Exclusion Criteria:

* Those in whom the total serum bilirubin (TSB) level rose by more than 5 mg/dl per day or was higher than 20 mg/dl within the first 24 hours after birth were excluded from the study.
* Infant of diabetic mothers.
* Maternal eclampsia-preeclampsia.
* Birth asphyxia
* Sepsis
* congenital anomalies.
* Direct Coombs'test positive
* Pathological causes of hyperbilirubinemia.
* Enclosed hemorrhage.
* Hemolytic type of hyperbilirubinemia due to blood group or Rh incompatibility.

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Effect of types of phototherapy on change in total antioxidant capacity (TAC) | 2 days
  This will be determined by:
  1. Measure TAC (mmol/L) before and after phototherapy
  2. Compare results of TAC (mmol/L) before and after phototherapy.
Effect of types of phototherapy on change in malonaldehyde (MDA) | 2 days
  This will be determined by:
  1. Measure MDA (nmol/L) before and after phototherapy
  2. Compare results of MDA (nmol/L) before and after phototherapy.
Effect of types of phototherapy on change in nitric oxide (NO) | 2 days
  This will be determined by:
  1. Measure NO (umol/L) before and after phototherapy
  2. Compare results of NO (umol/L) before and after phototherapy.

SECONDARY OUTCOMES:
Effect of types of phototherapy on change in serum iron (Fe) | 2 days
  This will be determined by:
  1. Measure serum Fe before and after phototherapy
  2. Compare results of serum Fe before and after phototherapy.
Effect of types of phototherapy on change in serum copper (Cu) | 2 days
  This will be determined by:
  1. Measure serum Cu before and after phototherapy
  2. Compare results of serum Cu before and after phototherapy.
Effect of types of phototherapy on change in serum zinc (Zn) | 2 days
  This will be determined by:
  1. Measure serum Zn before and after phototherapy
  2. Compare results of serum Zn before and after phototherapy.
Effect of types of phototherapy on change in serum calcium (Zn) | 2 days
  This will be determined by:
  1. Measure serum Ca before and after phototherapy
  2. Compare results of serum Ca before and after phototherapy.

REFERENCES:
- [Derived] El-Farrash RA, El-Shimy MS, Tawfik S, Nada AS, Salem DAD, M Gallo MS, Abd-Elmohsen EW. Effect of phototherapy on oxidant/antioxidant status: a randomized controlled trial. Free Radic Res. 2019 Feb;53(2):179-186. doi: 10.1080/10715762.2018.1549364. Epub 2019 Mar 1. PMID 30458636